CLINICAL TRIAL: NCT06886672
Title: Genetic Susceptibility in MAlignant Pleural Mesothelioma: Clinical Implication of GermliNE VariaTionS
Acronym: MAGNETS
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Istituti Clinici Scientifici Maugeri di Pavia (Unknown)
Responsible Party: Principal Investigator, Giulia Maria Stella, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: MAGNETS
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Mesothelioma, Malignant Pleural
Keywords: MPM; germline mutations; asbestos exposure
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: patients affected by MPM
- Cohort B: asbestos exposed subjects

SUMMARY:
Malignant pleural mesothelioma (MPM) is a rare and aggressive neoplasm of the pleural mesothelium, mainly associated to asbestos exposure, still lacking effective therapies.

Asbestos is a not-mutagenic agent: its nanosized fibres directly interact with tyrosine kinases (TKs) (e.g. EGFR) and may induce inappropriate receptor dimerization and activation, in absence of activating somatic mutations. TK receptor activation initiates cell signaling cascades and carcinogenesis. Asbestos, thus, induces the generation of an inflammatory immunosuppressive microenvironment that may support tumor growth in individuals with genetic predisposition (2). Consequently, the lack of actionable tumor targets together with the heterogeneous stroma, support the failure of modern drugs, both TK and immune-checkpoint inhibitors (TKIs, ICIs). In this complex context, the role of germline changes in MPM remains largely unexplored, except for changes in the BAP1 gene which are known to predispose to the disease (3).

The main goal of the study is to look for germline changes of a panel of genes involved in microenvironment infiltration modulation, drug response and cancer predisposition. The study will be performed in parallel on blood samples obtained from asbestos-exposed subjects and on MPM patients. This approach will allow: detection of putative germline signatures associated with MPM onset predisposition (or even protection) with prognostic and predictive implications.

The genetic characterization of MPM has not been fully clarified until now due to the significant inter-patient variability and to the scarcely reported somatic aberrations. Most of genetic alterations in MPM are loss of function of tumor suppressor genes or caretaker genes. Thus, the present project aimed at deeply investigate the germline variation in MPM and exposed population to determine host factors involved in MPM promotion. Pathogenic germline variants in MPM are often involved in DNA damage repair and chromatin remodeling pathways, and the most frequently identified germline mutations are in BAP1 which encodes for a tumor suppressor gene. Its protein is a nuclear deubiquitinating enzyme that plays an important role in chromatin modulation, transcriptional regulation, cell proliferation, DNA repair, cell death, and glucidic metabolism.

Based on systematic literature review performed to identify all relevant data, a set of 30 genes involved in microenvironment infiltration modulation (e.g. RBL1), drug response (e.g. XRCC1) and cancer predisposition (e.g. BRAC1-2) has been defined. This phase will encompass a first step focused on deep mutational screening aimed at analyzing a custom panel of genes involved in microenvironment immune-inflammatory on peripheral blood mononuclear cell (PBMC)-derived DNA. A next-generation sequencing (NGS) approach will be applied by Illumina-iSeq 100 Sequencing System. From each subject enrolled in this study, total DNA will be extracted by automated purification system, then 20 ng of input DNA will be used for library construction and next generation sequencing of all coding exons from cancer related gene. The identified variants will be submitted to bioinformatics analysis by PolyPhen-2, SIFT and Ensembl Variant Effect Predictor (VEP), to assess the possible impact of the corresponding amino acid substitution on the structure and function of the encoded protein. In addition, clinically significant variants will be annotated by using ClinVar-NCBI, GnomAD and COSMIC databases. Recent clinical studies have associated high tumor mutational burden (TMB) with improved patient response rates and survival benefit from immune checkpoint inhibitors; hence, TMB is emerging as a biomarker of response for these immunotherapy agents. Moreover, it has been shown that germline variants can influence the molecular phenotypes of tumors and thus predict the checkpoint inhibitors efficacy. Staring from these considerations, in this study we will also analyze the germline tumor mutational burden (gTMB) by assessing the total number of nonsynonymous mutations in each selected gene.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a rare and aggressive neoplasm of the pleural mesothelium, mainly associated to asbestos exposure, still lacking effective therapies. Incidence rates in Europe are projected to peak around 2025, due to the long latency between exposure and disease onset. Asbestos industrial use was at its peak in the 1970s and ceased in Italy in 1994 (L.D. 257). However, in the Pavia province, reclamation of the cement plant in Broni town started in 2007: the works are not yet completed, and exposure of the population continues today. The network of ASST Pavia province and IRCCS Policlinico San Matteo Foundation identified more than 80 incident cases in the last 2 years. Therefore, we have drawn our attention to a rare cancer, with a low life expectancy (12-15 months from diagnosis). Other diseases, even with same embryologic origin from mesoderm, such as ovarian cancers, are more common, well studied and have more established therapies. We also feel the need to respond to the specific welfare and unmet needs of our territory. Inhaled asbestos fibers migrate to the pleura, where they persist, cause irritation, perpetuate tissue damage and can be found post-mortem (1).

Asbestos is a not-mutagenic agent: its nanosized fibres directly interact with tyrosine kinases (TKs) (e.g. EGFR) and may induce inappropriate receptor dimerization and activation, in absence of activating somatic mutations. TK receptor activation initiates cell signaling cascades and carcinogenesis. Asbestos, thus, induces the generation of an inflammatory immunosuppressive microenvironment that may support tumor growth in individuals with genetic predisposition (2). Consequently, the lack of actionable tumor targets together with the heterogeneous stroma, support the failure of modern drugs, both TK and immune-checkpoint inhibitors (TKIs, ICIs). In this complex context, the role of germline changes in MPM remains largely unexplored, except for changes in the BAP1 gene which are known to predispose to the disease (3).

We will focus on a panel of genes involved in inflammatory infiltration, drug response, cancer predisposition to define germline signatures with potential prognostic and predictive implications. This study will contribute to decipher a still unexplored milieu and improve mechanistic knowledge on MPM biology and interindividual susceptibility to asbestos. Moreover, it could be of help in identifying novel actionable targets and in designing personalized and more efficient therapeutic strategies.

The main goal of the study is to look for germline changes of a panel of genes involved in microenvironment infiltration modulation, drug response and cancer predisposition. The study will be performed in parallel on blood samples obtained from asbestos-exposed subjects and on MPM patients. This approach will allow: i) detection of putative germline signatures associated with MPM onset predisposition (or even protection) with prognostic and predictive implications.

Primary aim will be the comparison of prevalence of germline mutations in MPM patients vs asbestos exposed healthy subjects.

Secondary aim will be the comparison of overall survival (OS) according to mutational status in MPM patients.

The study will be structured on three phases. The first step will regard sample collection. Patients affected by MPM, followed in the Pneumology Unit will be candidate to the study (30 cases/year).

For each of them a 4mL whole blood will be collected by blood draw (using EDTA as anticoagulant). Comparable quantity of blood will be derived from the biobank already viable at ICS Maugeri obtained from MPM patients (50 cases) and asbestos exposed subjects (30 cases). The oncological biobanks service unit is located at research laboratories of ICS Maugeri. It was funded in 2009 aimed at the collection, conservation, storage, and distribution of human biological material for research purposes. In the Maugeri institutional oncological biobank, biological samples from patients suffering from different types of cancer have been stored to date (4% malignant pleural mesothelioma) and for which clinical history and follow-up are well documented. For each enrolled case, clinical and demographic data will be collected by the PI after obtained a written informed consent. MPM patients will be treated according to international guidelines and managed based on the Interdisciplinary Group for Thoracic Neoplasms (GINT) evaluation.

The next step of the project encompasses a comprehensive and in-depth discovery effort aimed at identifying germline variations affecting a panel of genes involved in microenvironmental infiltrate regulation, drug response, and cancer susceptibility. Characterization of tumors utilizing next-generation sequencing methods is currently at the forefront of the field of personalized medicine. It should be underlined that in most cancer types, the genetic asset should be defined as a landscape consisting of a small number of mountains (genes altered in a high percentage of tumors) and a much larger number of hills, namely those genes altered infrequently. Published studies have revealed about 140 genes that, when altered by intragenic mutations, can promote or drive tumorigenesis; other mutations are passengers and do not confer elective growth advantage. On the other hand, several genes are known to predispose to cancer when inherited in mutant form in the germ line and are not somatically mutated in cancer to a substantial degree. These genes do not confer a significant selective growth advantage when changed but can promote tumorigenesis in indirect ways. The genetic characterization of MPM has not been fully clarified until now due to the significant inter-patient variability and to the scarcely reported somatic aberrations. Most of genetic alterations in MPM are loss of function of tumor suppressor genes or caretaker genes. In absence of a context of oncogenic addiction, pharmaceutical targeting of activated transducers (mTor inhibitors, FAK inhibitors) might hold a key to improve MPM therapy. Thus, the present project aimed at deeply investigate the germline variation in MPM and exposed population to determine host factors involved in MPM promotion. Pathogenic germline variants in MPM are often involved in DNA damage repair and chromatin remodeling pathways, and the most frequently identified germline mutations are in BAP1 which encodes for a tumor suppressor gene. Its protein is a nuclear deubiquitinating enzyme that plays an important role in chromatin modulation, transcriptional regulation, cell proliferation, DNA repair, cell death, and glucidic metabolism.

Based on systematic literature review performed to identify all relevant data, a set of 30 genes involved in microenvironment infiltration modulation (e.g. RBL1), drug response (e.g. XRCC1) and cancer predisposition (e.g. BRAC1-2) has been defined. This phase will encompass a first step focused on deep mutational screening aimed at analyzing a custom panel of genes involved in microenvironment immune-inflammatory on peripheral blood mononuclear cell (PBMC)-derived DNA. A next-generation sequencing (NGS) approach will be applied by Illumina-iSeq 100 Sequencing System. From each subject enrolled in this study, total DNA will be extracted by automated purification system, then 20 ng of input DNA will be used for library construction and next generation sequencing of all coding exons from cancer related gene. The identified variants will be submitted to bioinformatics analysis by PolyPhen-2, SIFT and Ensembl Variant Effect Predictor (VEP), to assess the possible impact of the corresponding amino acid substitution on the structure and function of the encoded protein. In addition, clinically significant variants will be annotated by using ClinVar-NCBI, GnomAD and COSMIC databases. Recent clinical studies have associated high tumor mutational burden (TMB) with improved patient response rates and survival benefit from immune checkpoint inhibitors; hence, TMB is emerging as a biomarker of response for these immunotherapy agents. Moreover, it has been shown that germline variants can influence the molecular phenotypes of tumors and thus predict the checkpoint inhibitors efficacy. Staring from these considerations, in this study we will also analyze the germline tumor mutational burden (gTMB) by assessing the total number of nonsynonymous mutations in each selected gene.

ELIGIBILITY:
Inclusion Criteria Cohort A:

* Patient with a documented diagnosis of MPM (any disease stage and independently from chemo line treatment)
* Age ≥ 18 years (there is no upper age limit).
* Patient who gives their informed consent to participate in the study

Exclusion Criteria Cohort A:

* No exclusion criteria

Inclusion Criteria Cohort B:

* Former asbestos exposed healthy subjects
* Age ≥ 18 years (there is no upper age limit).
* Subject who gives their informed consent to participate in the study

Exclusion Criteria Cohort B:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two different study populations will be candidate to the study:
  Cohort A- patients affected by MPM, followed in the Pneumology Units (IRCCS Policlinico San Matteo Foundation and Oncology Unit at ICS Maugeri IRCCS); Cohort B- asbestos exposed subjects, followed in the Occupational Hospital Medicine Unit (UOOML) at ICS Maugeri IRCCS.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the comparison of prevalence of germline mutations in MPM patients vs asbestos exposed healthy subjects | At enrollment visit 4mL whole blood will be collected by blood draw
  From each subject enrolled, DNA will be extracted by automated purification system. 20ng of input DNA will be used for library construction and next generation sequencing of all coding exons from cancer related gene. The identified variants will be submitted to bioinformatics analysis by PolyPhen-2, SIFT and Ensembl Variant Effect Predictor, to assess the possible impact of the corresponding amino acid substitution on structure and function of the encoded protein. Clinically significant variants will be annotated using ClinVar-NCBI, GnomAD, COSMIC databases. Recent studies have associated high tumor mutational burden with improved patient response rates and survival benefit from immune checkpoint inhibitors. It has been shown that germline variants can influence the molecular phenotypes of tumors and thus predict the checkpoint inhibitors efficacy. We will analyze the germline tumor mutational burden by assessing the total number of nonsynonymous mutations in each selected gene.

SECONDARY OUTCOMES:
Secondary aim will be the comparison of overall survival (OS) according to mutational status in MPM patients. | From enrollment until 12 months, or until the participant is lost to follow-up
  Participants will undergo the following evaluations at baseline: clinical and demographic data, concurrent medication, comorbidities, smoking habits, occupational exposure and genetic evaluation from whole blood sample.
  Clinically changes will be followed until 12 months, or until the participant is lost to follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - IRCCS Istituti Clinici Maugeri, Medicina del Lavoro, Pavia, Pavia

REFERENCES:
- [Background] Testa JR, Cheung M, Pei J, Below JE, Tan Y, Sementino E, Cox NJ, Dogan AU, Pass HI, Trusa S, Hesdorffer M, Nasu M, Powers A, Rivera Z, Comertpay S, Tanji M, Gaudino G, Yang H, Carbone M. Germline BAP1 mutations predispose to malignant mesothelioma. Nat Genet. 2011 Aug 28;43(10):1022-5. doi: 10.1038/ng.912. PMID 21874000
- [Background] Lettieri S, Bortolotto C, Agustoni F, Lococo F, Lancia A, Comoli P, Corsico AG, Stella GM. The Evolving Landscape of the Molecular Epidemiology of Malignant Pleural Mesothelioma. J Clin Med. 2021 Mar 3;10(5):1034. doi: 10.3390/jcm10051034. PMID 33802313
- [Background] Roe OD, Stella GM. Malignant pleural mesothelioma: history, controversy and future of a manmade epidemic. Eur Respir Rev. 2015 Mar;24(135):115-31. doi: 10.1183/09059180.00007014. PMID 25726562